CLINICAL TRIAL: NCT06807216
Title: Feasibility Study Assessing Content and Delivery of the YATAC Programme
Brief Title: Evaluating Feasibility of the YATAC Programme
Acronym: YATAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Defactum, Central Denmark Region (Other Government)
Collaborators: Gødstrup Hospital (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Marc Sampedro Pilegaard, Senior Researcher and Associate Professor, Defactum, Central Denmark Region
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: S-20240101
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: Feasibility; Rehabilitation; young adults; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A repeated-measurement one-armed feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YATAC (Experimental): The programme draws on a person-centered approach and is designed to enhance the constructs of social cognitive theory, with an emphasis on self-efficacy .The programme comprises seven components, with several sessions providing knowledge, strategies, and practical exercises. The intervention starts with one mandatory component: 1) needs assessment and goal setting. These inform which, when, and how many sessions within the following components the participants will receive:
  2. Everyday life 3. Physical activity 4. Psychological issues 5. Education and work 6. Sexuality and relationship 7. Family and friends
  The programme is delivered over 16 weeks, primarily as a group-based intervention. The components last 30-120 minutes and are provided by an interdisciplinary team at rehabilitation centers.
  Interventions: Behavioral: YATAC

INTERVENTIONS:
Behavioral: YATAC — Age-specific rehabilitation for young adult cancer survivors

SUMMARY:
Between 2019 and 2023, the Young Adult Taking Action (YATAC) program was developed to support young adults recovering from cancer. The program is based on three key studies:

* A review of previous programs designed to help young adult cancer survivors.
* A study where young adults, their families and friends, and healthcare professionals shared what kind of support young people need to return to everyday life.
* A collaborative process where young adults, professionals, and researchers worked together to design the program's content and how it should be delivered.

YATAC is specifically designed for young adults and includes different areas of support, such as setting goals, managing daily life, staying active, coping with psychological challenges, navigating education and work, understanding rights and finances, relationships and sexuality, family and friends, and peer-to-peer support.

The first phase of the project was funded by the Danish Cancer Society, the Region of Southern Denmark, the University of Southern Denmark, and REHPA, the Danish Knowledge Centre for Rehabilitation and Palliative Care.

One of the study in the second phase includes:

Study 1: A feasibility study to see if young adults find the program relevant and helpful, and whether they are able to participate. A total of 40 young adults will try the program at the Center for Cancer and Health in Copenhagen. The findings will help refine the program so it can be adapted to local healthcare services.

The results from these studies will provide valuable insights into how to better support young adult cancer survivors and reduce the long-term challenges they face. The program is expected to improve their quality of life while also helping to reduce healthcare costs and social inequality.

DETAILED DESCRIPTION:
Young adult cancer survivors aged 18-39 experience extensive age-specific late effects after cancer treatment affecting their everyday life; yet, they are not receiving rehabilitation after ending treatment, leading to reduced health-related quality of life (HRQoL).

In 2019, the 'Young Adult Taking Action' (YATAC) programme was established to develop a rehabilitation programme supporting young adult cancer survivors in taking control over their everyday life and increasing their HRQoL. The programme is a person-centred, goal-oriented, interdisciplinary and peer-based intervention. It is delivered over 16 weeks, primarily as a group-based intervention and consists of the following components:

1. Needs assessment and goal setting
2. Everyday life
3. Physical activity
4. Mental health
5. Education and work
6. Sexuality and relationship
7. Family and friends

The overall perspectives are to improve quality of life, self-efficacy, functioning and reduce cancer and treatment-related late effects in young adult cancer survivors.

The programme has undergone a development process and is now ready to be tested to prepare national scalability.

The study include:

1) A feasibility study assessing the content and delivery of the YATAC programme for young adult cancer survivors in the Municipality of Copenhagen. Qualitative and quantitative data will be collected about acceptability of the programme and its intervention components, potential mechanisms of action, perceived value, benefits, harms, and unintended consequences and fidelity, reach, and dose. Furthermore, costs related to content and delivery of the YATAC programme will also be evaluated.

The project will potentially change rehabilitation practice in Danish municipalities for young adult cancer survivors and reduce the disabling late effects from cancer treatment, so they can obtain the best possible HRQoL.

ELIGIBILITY:
Inclusion Criteria:

* Included participants will be between 18-39 years old with any cancer diagnosis,
* Undergoing or having undergone curative intended cancer treatment
* Reporting a rehabilitation need
* Speaking and understanding the Danish language
* Living in the Municipality of Copenhagen

Exclusion Criteria:

* Young people aged 18-39 who were diagnosed with cancer before the age of 18.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Quantitative data | Qualitative will be collected during the 16 weeks of intervention, including baseline (T1), session delivery (T2), and the end of the 16 weeks (T3).
  Quantitative data from professionals delivering the programme: Paper-based forms will collect data about fidelity, dose, and the programme's overall value.
  Quantitative data from participants: They will report their perceived value of each session, the degree to which they could participate in each session, the overall value of the programme regarding improvement in everyday life and self-efficacy, and the degree to which they have adopted the content from the sessions into their everyday lives. Furthermore, the investigators will also evaluate the value of using peer-to-peer support.

SECONDARY OUTCOMES:
Qualitative data | End at 16 weeks
  Qualitative data from participants: A purposively selected sample of the participants will be invited to participate in a semi-structured focus group interview focusing on perceived benefits, harms, unintended consequences, and acceptability (n=10).
  Qualitative data from professionals: The professionals will be invited to a focus group interview on the same aspects as above.

OTHER OUTCOMES:
Costs | Baseline, during delivery and end of programme at 16 weeks.
  Resource use associated with programme delivery will be tested to ensure high-quality measurements, enabling the following cost estimation for the intervention. Moreover, a costing questionnaire registering background information, health service use and productivity loss will be tested among the participants to enable a future cost-effectiveness analysis of the YATAC programme.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Center for Kræft og Sundhed, Copenhagen, København N
  - Center for Kræft og Sundhed, Copenhagen N

IPD SHARING:
Plan to Share IPD: No